CLINICAL TRIAL: NCT01634568
Title: A Double-blind, Randomised, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of V81444 in Healthy Male Volunteers
Brief Title: A Clinical Trial to Find Out V81444's Side Effects and Blood Levels in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: V81444-1PD-01; 2011-001975-38 (EudraCT Number)
Record Dates: First submitted 2012-06-20; First posted 2012-07-06 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Ascending Dose (Experimental): Single Ascending Doses of V81444 compared to placebo
  Interventions: Drug: V81444
- Multiple Ascending Doses (Experimental): Multiple ascending doses of V81444 compared to placebo
  Interventions: Drug: V81444

INTERVENTIONS:
Drug: V81444 — Single ascending oral doses of V81444 and placebo
  Multiple ascending oral doses of V81444 and placebo

SUMMARY:
A double-blind, randomised, placebo-controlled study of the safety, tolerability and pharmacokinetics of single and multiple ascending oral doses of V81444 in healthy male volunteers

DETAILED DESCRIPTION:
Part A - Single Ascending Dose (SAD) Double-blind, randomised, placebo-controlled, single ascending dose study.

Each study subject will participate in a screen visit, three identical treatment periods, in each of which they will receive a single oral dose of V81444 or placebo in accord-ance with the randomisation schedule, and one post-study visit.

In each treatment period, subjects will be admitted the day before dosing (Day -1) and, subject to satisfactory medical review, discharged in the morning, 4 days later (Day 4).

Part B - Multiple Ascending Dose (MAD) Double-blind, randomised, placebo-controlled, parallel group, multiple ascending dose study

Each study subject will participate in a screen visit, one treatment period in which they will receive repeated oral doses of V81444 or placebo in accordance with the randomisation schedule, and one post-study visit.

In each treatment period, subjects will be admitted the day before dosing (Day -1), dosed daily on Days 1 to 14 and, subject to satisfactory medical review, will be discharged in the morning, 3 days after the final dose (Day 17).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers: aged 18 to 45 years, in good general health as determined by medical history, physical examination and screening investigations, and taking no regular medication. Confirmation to be sought for all volunteers that their general practitioner has provided an acceptable medical history.

Exclusion Criteria:

* have a history or evidence of clinically significant gastrointestinal disease, including ulcers, gastro-oesophageal reflux disease or gastritis
* any known malformations that would make OGD difficult or unsafe(Part B only)
* have taken V81444 in any previous investigational study
* have taken any restricted concomitant medication
* have multiple drug allergies or be allergic to any of the components of V81444 study medication or its matching placebo or midazolam (Part B only)
* in the 4 calendar months before study drug administration have smoked more than 5 cigarettes per day have consumed more than 28 units of alcohol per week have donated blood or plasma in excess of 500 mL been exposed to any new investigational agent or any other adenosine A2A receptor antagonist used non-steroidal anti-inflammatory drugs regularly had a new tattoo or body piercing
* have any clinically relevant abnormal findings at screening and/or admission
* intend to father a child with their female partner or through sperm donation within 4 months after the last dose of study medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of V81444 by assessing the frequency of adverse events | From screening until 7 days post dosing
Evaluate the safety of V81444 by assessing laboratory safety assessments | Lab safety assessments are taken at screening, day minus 1, 24h and 72h and post dosing
Evaluate the safety of V81444 by assessing ECG | Taken at screening and until 7 days post dosing
Evaluate the safety of V81444 by assessing vital signs | Taken at screening and until 7 days post dosing
Evaluate the safety of V81444 by assessing physical examination | Taken at screening and post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Steve Warrington, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom